CLINICAL TRIAL: NCT01479699
Title: Absorption and Metabolism of Olive Leaf Extract and Its Effect on Vascular Reactivity and Cytokine Concentrations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Comvita UK (Unknown)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Professor of Biochemistry, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: OLE study
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Absorption and Metabolism; Effect on Vascular Function; Effect on Cytokine Concentrations
Keywords: Olive leaf extract; Polyphenols; Vascular function; Bioavailability; Cytokines
MeSH Terms: interventions — olive leaf extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo capsule (Placebo Comparator): Four placebo capsules containing safflower oil only
  Interventions: Dietary Supplement: Olive leaf extract capsules
- Olive leaf extract capsule (Active Comparator): Four olive leaf capsules. Each containing 4mg oleuropein plus safflower oil.
  Interventions: Dietary Supplement: Olive leaf extract capsules

INTERVENTIONS:
Dietary Supplement: Olive leaf extract capsules — Four capsules taken at baseline each containing 4mg oleuropein

SUMMARY:
The purpose of this study is to determine how olive leaf is absorbed and metabolised and also whether it has any effect on the elasticity of blood vessels and the immune system.

DETAILED DESCRIPTION:
The purpose of this study is to determine how olive leaf is absorbed and metabolised and also whether it has any effect on vascular function and cytokine concentrations.

ELIGIBILITY:
Inclusion Criteria:

* 19-40 years, non-smokers, able to swallow capsules, have a Body Mass Index (BMI) of 18.5-30, have a normal liver function and haematology and a max alcohol intake of <21 units/week

Exclusion Criteria:

* Those who suffer from any form of disease, including endocrine disease, liver disease, diabetes mellitus, myocardial infarction, blood clotting disorder, reproductive disorder, gastrointestinal disease or a chronic gastrointestinal disorder.
* Individuals who are vegetarian, have dietary restrictions or on a weight reducing diet will not be recruited.
* Subjects who have been taking antibiotics in previous 3 months before study will not be included in the study
* Females who may be pregnant, or if of childbearing potential and are not using effective contraceptive precautions will be excluded.
* Blood pressure > 150/90 mmHg
* Haemoglobin < 125 g/l for male, < 110 g/l for female
* Gamma GT (liver enzymes) > 80 IU/l
* Cholesterol > 6.5 mmol/l
* Had suffered a myocardial infarction or stroke in the previous 12 months
* On any lipid-modifying medication
* On any medication affecting blood clotting
* Individuals taking vitamin and/or fish oil supplements

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Absorption and metabolism | 0. 0.5, 1, 1.5, 2, 3, 4, 6, 8 hours post ingestion (blood) 0, 0-4, 4-8 and 8-24 hours post ingestion (urine)
  Olive leaf polyphenol metabolites measured in blood and urine samples

SECONDARY OUTCOMES:
Vascular function | 0, 2, 4, 6 hours post ingestion (LDI) 0, 0.5, 1, 1.5, 2, 3, 4, 6 and 8 hours post ingestion (DVP)
  Vascular function was assessed via two methods: Laser Doppler Iontophoresis (LDI) and Digital Volume Pulse (DVP)
Cytokine concentration | 0, 1, 3 and 6 hours post ingestion
  Concentrations of IL-8, IL-1beta, IL-6, IL-10 and TNF-alpha will be measured in whole blood stimulated with LPS.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy PE Spencer, PhD, Principal Investigator — University of Reading; Ian Rowland, PhD, Principal Investigator — University of Reading; Parveen Yaqoob, PhD, Principal Investigator — University of Reading
Locations (1):
- Hugh Sinclair Unit of Human Nutrition, University of Reading, Reading, Berkshire, United Kingdom